CLINICAL TRIAL: NCT03537430
Title: Totally no Tube (TNT) Uniportal Video-assisted Thoracoscopic Surgery (VATS) VS Traditional Uniportal VATS for Mediastinal Tumor: A Prospective Randomized Controlled Trial
Brief Title: Totally no Tube (TNT) Uniportal Video-assisted Thoracoscopic Surgery (VATS) VS Traditional Uniportal VATS for Mediastinal Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xueying Yang (Other)
Responsible Party: Sponsor-Investigator, Xueying Yang, Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC-2018-HS-001
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Mediastinal Tumor
Keywords: TNT (Totally no tube); uniportal VATS; mediastinal tumor
MeSH Terms: conditions — Mediastinal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-center prospective randomized controlled trial. 98 patients aged between 18 and 75 years with clinically mediastinal tumors were randomly assigned to two groups, 50 patients received TNT uniportal VATS mediastinal tumor resection (TNT group) and 48 patients underwent traditional uniportal VATS mediastinal tumor resection (control group), the short-term perioperative outcomes would be reported here.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: This study is a prospective randomized controlled clinical trial. Participants, care provider, and investigator all know the grouping situation. The Investigator collect the information and observation indicators of the two groups of participants and send to the Outcomes Assessor . The Outcomes Assessor does not know the grouping situation of each participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNT Uniportal Video-assisted Thoracoscopic Surgery (Other): This group of patients underwent TNT uniportal VATS mediastinal tumor resection
  Interventions: Procedure: TNT uniportal VATS mediastinal tumor resection
- Uniportal Video-assisted Thoracoscopic Surgery (Other): This group of patients underwent traditional uniportal VATS mediastinal tumor resection
  Interventions: Procedure: Traditional uniportal VATS mediastinal tumor resection

INTERVENTIONS:
Procedure: TNT uniportal VATS mediastinal tumor resection — TNT uniportal video-assisted thoracoscopic surgery refers to the use of conventional uniportal video-assisted thoracoscopic surgery, the use of laryngeal mask anesthesia instead of tracheal intubation anesthesia, intraoperative catheter was not retained, postoperative chest catheter placement.
  Arms: TNT Uniportal Video-assisted Thoracoscopic Surgery
Procedure: Traditional uniportal VATS mediastinal tumor resection — The surgical procedures followed principles of mediastinal tumor resection，uniportal video-assisted thoracoscopic surgery in mediastinal tumor resection.
  Arms: Uniportal Video-assisted Thoracoscopic Surgery

SUMMARY:
TNT surgery is a new area of exploration and evolution in thoracic minimal invasive surgery. TNT Uniportal Video-assisted Thoracoscopic Surgery (VATS) has become popular during mediastinal tumors resection. However, there has been little randomized controlled trials into the associated feasibility and advantage. The aim of our RCT was to evaluate the feasibility and advantage of TNT Uniportal VATS for mediastinal tumors resection and its significance in Fast Track Surgery (FTS). This is a single-center prospective randomized controlled trial. 98 patients aged between 18 and 75 years with clinically mediastinal tumors were randomly assigned to two groups, 50 patients received TNT uniportal VATS mediastinal tumor resection (TNT group) and 48 patients underwent traditional uniportal VATS mediastinal tumor resection (control group), the short-term perioperative outcomes would be reported here.

DETAILED DESCRIPTION:
This study was designed as a single-center prospective randomized controlled trial. The trial recruited patients aged from 18 to 75 years with a diagnosis of mediastinal tumor. Preoperative chest CT examination showed that shape of the mediastinal tumor was regular, boundary was clear, and maximum diameter of the mass was less than 4 cm. Other inclusion criteria included capability of giving consent and adequate organ function to tolerate uniportal thoracoscopy mediastinal tumor resection. The exclusion criteria are described as follows: preoperative examination showed that the tumor invaded the surrounding blood vessels, pericardium, lung and other tissues or had distant metastasis; preoperative complications include severe coronary heart disease, arrhythmia and other serious cardiopulmonary diseases; large masses, difficult surgical procedures; manifestations of myasthenia gravis; hypovolemia, blood disorders, or abnormal clotting mechanism; pulmonary function and arterial blood gas analysis showed that patients could not tolerate surgery; previous thoracotomy; inability to obtain consent. Furthermore, the exclusion criteria were defifined as follows: intraoperative pleural adhesion or technical challenge to achieve hemostasis that make conversion from VATS to thoracotomy; clinician decides the patient should not continue the trial according to individual condition; patient withdraws from the trial. According to International Conference on Harmonisation, all participants gave written informed consent. Our RCT was launched in April 2018, which conducted in accordance with the Declaration of Helsinki and good clinical practice according to the International Conference on Harmonization guidelines. The ethics committee of The Fourth Affiliated Hospital of Medical Sciences, Liaoning, China, approved this study (approval number: EC-2018-HS-01).

After eligibility had been confirmed and inform consents obtained, the investigator registered patients to ensure allocation concealment. Next we randomly enrolled patients to TNT group and control group in accordance with a list of randomization numbers. This list was generated in the trial statistician's computer. Allocation was communicated by telephone by the trial coordinator. Neither patients nor any investigators were masked to treatment allocation.

The patients underwent routine physical examination, hematologic and biochemical tests, arterial blood gas analysis, pulmonary function test and computed tomography. Uniportal VATS mediastinal tumor resection was the standard surgical intervention according to the protocol. Patients in TNT group underwent TNT uniportal VATS mediastinal tumor resection, patients in control group underwent traditional uniportal VATS. Pre-, peri-, and postoperative details and outcome variables of patients were collected.

ELIGIBILITY:
Inclusion Criteria:

The trial recruited patients aged from 18 to 75 years with a diagnosis of mediastinal tumor. Preoperative chest CT examination showed that shape of the mediastinal tumor was regular, boundary was clear, and maximum diameter of the mass was less than 4 cm. Other inclusion criteria included capability of giving consent and adequate organ function to tolerate uniportal thoracoscopy mediastinal tumor resection.

Exclusion Criteria:

Preoperative examination showed that the tumor invaded the surrounding blood vessels, pericardium, lung and other tissues or had distant metastasis; preoperative complications include severe coronary heart disease, arrhythmia and other serious cardiopulmonary diseases; large masses, difficult surgical procedures; manifestations of myasthenia gravis; hypovolemia, blood disorders, or abnormal clotting mechanism; pulmonary function and arterial blood gas analysis showed that patients could not tolerate surgery; previous thoracotomy; inability to obtain consent. Furthermore, the exclusion criteria were defifined as follows: intraoperative pleural adhesion or technical challenge to achieve hemostasis that make conversion from VATS to thoracotomy; clinician decides the patient should not continue the trial according to individual condition; patient withdraws from the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
operative time | 1 day
  Anesthesia completed to the end of the operation
Intubation/laryngeal mask completion time | 1 day
  Intubation/laryngeal mask completion time
duration of postoperative pain | 10 days
  Postoperative pain duration
VAS pain scores | 5 days
  The VAS pain score was given to patients and the pain scores were recorded at 6h, 12h, 24h, 48h, and 72h postoperatively.
Intraoperative blood loss | 1 day
  Intraoperative blood loss
The time of early ambulation after operation | 1 day
  The time from the patient's postoperative pushback to the first bedtime
Postoperative hospital stay | 15 days
  Postoperative hospital stay
hospitalization expenses | 15 days
  The total cost of hospitalization
Intraoperative oxygen saturation, SpO2 | 1 day
  Intraoperative oxygen saturation, SpO2
Intraoperative mean arterial pressure, MAP | 1 day
  Intraoperative mean arterial pressure, MAP
postoperative complication rate | 15 days
  Incidence of postoperative complications such as respiratory, cardiovascular and intubation-related complications
Intraoperative heart rate, HR | 1 day
  Intraoperative heart rate, HR
Postoperative extubation time | 1 day
  Postoperative extubation time
Postoperative feeding time | 1 day
  Postoperative feeding time

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Affiliated Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Result] Zhao ZR, Lau RWH, Ng CSH. Anaesthesiology for uniportal VATS: double lumen, single lumen and tubeless. J Vis Surg. 2017 Aug 21;3:108. doi: 10.21037/jovs.2017.07.05. eCollection 2017. PMID 29078668
- [Result] Petersen RH, Holbek BL, Hansen HJ, Kehlet H. Video-assisted thoracoscopic surgery-taking a step into the future. Eur J Cardiothorac Surg. 2017 Apr 1;51(4):694-695. doi: 10.1093/ejcts/ezw381. No abstract available. PMID 28007878
- [Result] Mineo TC, Tamburrini A, Perroni G, Ambrogi V. 1000 cases of tubeless video-assisted thoracic surgery at the Rome Tor Vergata University. Future Oncol. 2016 Dec;12(23s):13-18. doi: 10.2217/fon-2016-0348. Epub 2016 Sep 30. PMID 27686131
- [Result] Cui F, Liu J, Li S, Yin W, Xin X, Shao W, He J. Tubeless video-assisted thoracoscopic surgery (VATS) under non-intubated, intravenous anesthesia with spontaneous ventilation and no placement of chest tube postoperatively. J Thorac Dis. 2016 Aug;8(8):2226-32. doi: 10.21037/jtd.2016.08.02. PMID 27621880
- [Result] Gonzalez-Rivas D, Yang Y, Guido W, Jiang G. Non-intubated (tubeless) uniportal video-assisted thoracoscopic lobectomy. Ann Cardiothorac Surg. 2016 Mar;5(2):151-3. doi: 10.21037/acs.2016.03.02. No abstract available. PMID 27134844
- [Result] Fernandes P, Lareiro S, Vouga L, Guerra M, Miranda J. Uniportal Video-Assisted Thorascoscopic Surgery - The New Paradigm in the Surgical Treatment of Lung Cancer. Rev Port Cir Cardiotorac Vasc. 2017 Jul-Dec;24(3-4):127. PMID 29701369
- [Result] Migliore M. Uniportal video-assisted thoracic surgery, and the uni-surgeon: new words for the contemporary world. J Vis Surg. 2018 Mar 7;4:45. doi: 10.21037/jovs.2018.02.11. eCollection 2018. PMID 29682455
- [Result] Bedetti B, Solli P, Lawrence D, Panagiotopoulos N, Hayward M, Scarci M. Single port video-assisted thoracoscopic thymectomy. J Vis Surg. 2016 Sep 1;2:149. doi: 10.21037/jovs.2016.08.07. eCollection 2016. PMID 29078536
- [Result] Ooi A, Sibayan M. Uniportal video assisted thoracoscopic surgery thymectomy (right approach). J Vis Surg. 2016 Jan 17;2:13. doi: 10.3978/j.issn.2221-2965.2015.12.14. eCollection 2016. PMID 29078441
- [Result] Ooi A, Qiang F. Uniportal video assisted thoracoscopic surgery thymectomy (left approach). J Vis Surg. 2016 Jan 16;2:12. doi: 10.3978/j.issn.2221-2965.2015.12.18. eCollection 2016. PMID 29078440
- [Result] Dunning J. Video-assisted thoracoscopic microthymectomy. Ann Cardiothorac Surg. 2015 Nov;4(6):550-5. doi: 10.3978/j.issn.2225-319X.2015.11.04. PMID 26693152